CLINICAL TRIAL: NCT00555347
Title: Use of Armodafinil (R-modafinil) for Fatigue in Sarcoidosis
Brief Title: Use of Armodafinil for Fatigue in Sarcoidosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Principal Investigator, Robert P Baughman, Prof Medicine, University of Cincinnati
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB 07011901
Record Dates: First submitted 2007-11-07; First posted 2007-11-08 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2013-04

CONDITIONS: Sarcoidosis; Fatigue; Sleepiness
Keywords: Sarcoidosis; Fatigue
MeSH Terms: conditions — Sarcoidosis; Fatigue; Sleepiness | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Armnodafinil (Active Comparator): Armodafinil
  Interventions: Drug: Armodafinil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Armodafinil — Dosage 150-250 mg
  Other Names: Nuvigil
  Arms: Armnodafinil
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To determine the effect of Armodafinil (Nuvigil) on fatigue and sleep in sarcoidosis.

DETAILED DESCRIPTION:
The study will be divided into two halves. Patients will receive either drug or placebo in the first half. Patients receiving active drug will be started at one dose and it can be increased at the second visit. Those patients randomized to placebo will also have their dose adjusted by the investigating physician. The physicians will be blinded as to whether the patient is receiving drug or placebo. In the second half of the study, patients will receive the opposite treatment.

Patients will have complete detailed questionnaires regarding their fatigue, sleepiness, and overall quality of life.

They will have sleep studies done at the start and after each half of the study to determine the effect of therapy on sleepiness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sarcoidosis using standard criteria 15.
* Disease for more than one year
* On stable, systemic therapy
* Complain of fatigue which has been present for more than six months.
* Over 18 years of age
* Provide written informed consent.

Exclusion Criteria:

* Pregnancy
* Change in therapy for sarcoidosis in prior three months
* History of ventricular arrythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-10; Primary Completion 2010-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To determine the effect of Armodafinil (Nuvigil) on fatigue and sleep in sarcoidosis. | Prospective

SECONDARY OUTCOMES:
To determine the effect of Armodafinil (Nuvigil) on pulmonary function in sarcoidosis. | Prospective
To determine the safety and tolerability of Armodafinil (Nuvigil) in sarcoidosis. | Prospective

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Baughman, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States